CLINICAL TRIAL: NCT02058563
Title: Immunogenicity and Safety Study of GSK Biologicals' Combined Measles-mumps-rubella Vaccine in Subjects Seven Years and Older (209762)
Brief Title: Immunogenicity and Safety of GSK Biologicals' Combined Measles-mumps-rubella Vaccine in Volunteers, Seven Years of Age and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 115231; 2011-003672-36 (EudraCT Number)
Record Dates: First submitted 2014-02-06; First posted 2014-02-10 (Estimated); Results first posted 2017-04-10 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Rubella; Mumps; Measles
Keywords: Measles, mumps and rubella diseases; Safety; Immunogenicity
MeSH Terms: conditions — Rubella; Mumps; Measles | interventions — Measles-Mumps-Rubella Vaccine; Rubella Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- INV_MMR Group (Experimental): Subjects will receive 1 dose of GSK Biologicals' trivalent Measles, Mumps, and Rubella Virus Vaccine (Priorix®).
  Interventions: Biological: Priorix®
- COM_MMR Group (Active Comparator): Subjects will receive 1 dose of Merck's M-M-R®II, Measles, Mumps, and Rubella Virus Vaccine.
  Interventions: Biological: Merck's M-M-R®II, Measles, Mumps, and Rubella Virus Vaccine

INTERVENTIONS:
Biological: Priorix® — 1 dose administered as a subcutaneous (SC) injection.
  Arms: INV_MMR Group
Biological: Merck's M-M-R®II, Measles, Mumps, and Rubella Virus Vaccine — 1 dose administered subcutaneously.
  Arms: COM_MMR Group

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of GSK's trivalent MMR (Priorix®), comparing it to Merck"s MMR vaccine (M-M-R®II), which is approved for use in the US.

DETAILED DESCRIPTION:
This study will evaluate the immunogenicity of GSK's trivalent MMR vaccine (referred to as INV_MMR vaccine) in contrast to the US standard of care (M-M-R®II, Merck and Company, referred to as COM_MMR) when both are used as a second dose in subjects 7 years of age and older. In this study, the INV_MMR vaccine may be administered as a second dose to persons with either a history or formal documentation of at least one dose immunization with any MMR vaccine. This study is intended to support licensure of GSK's MMR vaccine in the US.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parent(s) or Legally Acceptable Representative(s) (LAR) can and will comply with the requirements of the protocol.
* Male or female subjects 7 years of age or older and born after December 31, 1956*. *The only exception to this is health care workers born before 1957 without other evidence of immunity to mumps for which one dose of a live mumps virus vaccine is recommended; therefore this population is eligible for enrollment in this study.
* For all children 7-17 years of age:

  * Written documentation of prior receipt of 1 dose of MMR vaccine administered on or after the first birthday.
* For all adults 18 years of age and older:

  * Prior receipt (written or verbal history) of at least one dose of MMR vaccine.
  * Birth in the US.
* Written informed consent obtained from the subject or from the parent(s)/LAR(s) of the subject (assent will be obtained from subjects who are still legally minors in line with local rules and regulations).
* Subjects in stable health as determined by investigator's physical examination and assessment of subjects' medical history.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, or ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject

  * Has agreed to be abstinent or practiced adequate contraception during the entire period starting 30 days prior to vaccination(s) until 3 months after receipt of the study vaccination and
  * has a negative pregnancy test on the day of vaccination.

Exclusion Criteria:

* Child in care.
* For all children 7-17 years of age:

  * Previous receipt of more than 1 dose of a measles-containing vaccine.
* Use of any investigational or non-registered product other than the study vaccine(s), during the period starting 30 days preceding the day of study vaccination, (i.e. 30 days prior to Day 0) or planned use during the entire study period.
* Receipt of any measles, mumps or rubella-containing vaccine during the period starting 42 days before the day of study vaccination (i.e. 42 days prior to Day 0).
* Chronic administration (defined as 14 or more consecutive days) of immunosuppressants or other immune-modifying drugs during the period starting 180 days before study vaccination or any planned administration of immune-modifying drugs during the entire study. Inhaled and topical steroids are allowed.
* Administration of immunoglobulins and/or any blood products during the period starting 180 days prior to study vaccination through the immunogenicity evaluation at Visit 2 or Visit 3 (for one-dose or two-dose cohort, respectively).
* Planned administration/ administration of any live viral vaccine not foreseen by the study protocol during the period starting 30 days prior to study vaccination and ending at Visit 2. Live intranasal influenza vaccine or any inactivated vaccine required in the age group may be given at any time, including the day of study vaccination.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* History of measles, mumps, or rubella disease.
* Known exposure to measles, mumps, or rubella, during the period starting 30 days before study start (i.e. 30 days prior to Day 0).
* %

Min Age: 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 996 (Actual)
Dates: Start 2014-07-01; Primary Completion 2015-05-24 (Actual); Study Completion 2015-09-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (16):
- United States (9):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Chandler, Arizona
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Edina, Minnesota
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, San Antonio, Texas
- GSK Investigational Site, Tartu, Estonia
- Slovakia (6):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Dolný Kubín
  - GSK Investigational Site, Dunajská Streda
  - GSK Investigational Site, Martin
  - GSK Investigational Site, Ružomberok
  - GSK Investigational Site, Zlaté Moravce

REFERENCES:
- [Derived] Abu-Elyazeed R, Jennings W, Severance R, Noss M, Caplanusi A, Povey M, Henry O. Immunogenicity and safety of a second dose of a measles-mumps-rubella vaccine administered to healthy participants 7 years of age or older: A phase III, randomized study. Hum Vaccin Immunother. 2018;14(11):2624-2631. doi: 10.1080/21645515.2018.1489186. Epub 2018 Jul 12. PMID 29902133

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 996 subjects were enrolled and 994 were vaccinated. Of the 994 vaccinated subjects, 83 subjects from 2 US sites were excluded due to significant GCP concerns, resulting in 911 subjects in the Total vaccinated cohort considered for the analysis.
Groups:
- INV_MMR Group: Subjects received one dose of INV_MMR (Priorix®) vaccine at Visit 1 (Day 0).
- COM_MMR Group: Subjects received one dose of COM_MMR (M-M-R®II ) vaccine from Lot 1 or Lot 2 at Visit 1 (Day 0).
Period: Overall Study
Arm/Group | INV_MMR Group | COM_MMR Group
Started | 454 | 457
Completed | 426 | 433
Not Completed | 28 | 24
Not completed — Lost to Follow-up | 26 | 22
Not completed — Other (vaccinated later as new subject) | 1 | 0
Not completed — Consent Withdrawal | 1 | 1
Not completed — Other (patient incarcerated) | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- COM_MMR Group: Subjects received one dose of COM_MMR (M-M-R®II) vaccine from Lot 1 or Lot 2 at Visit 1 (Day 0).
- Total: Total of all reporting groups
Arm/Group | INV_MMR Group | COM_MMR Group | Total
Number analyzed (Participants) | 454 | 457 | 911
Age, Continuous [Mean (Standard Deviation); unit: Months] | 25.9 (13.9) | 25.6 (13.8) | 25.7 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 250 | 252 | 502
  Male | 204 | 205 | 409
Race/Ethnicity, Customized [Number; unit: Participants]
  African Heritage/African American | 108 | 103 | 211
  American Indian or Alaskan native | 2 | 4 | 6
  Asian - Central/South Asian heritage | 1 | 0 | 1
  Asian - East Asian heritage | 1 | 0 | 1
  Asian - Japanese heritage | 0 | 1 | 1
  Asian - South East Asian heritage | 0 | 0 | 0
  Native Hawaiian or other Pacific Islander | 1 | 0 | 1
  White - Arabic/North African heritage | 0 | 1 | 1
  White - Caucasian/European heritage | 334 | 344 | 678
  Other | 7 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Anti-measles Virus Antibody Concentrations.
Description: Antibody concentrations are expressed as Geometric Mean Concentrations (GMCs) in milli International Units per milliliter (mIU/mL). Seropositivity was defined as subjects with anti-measles virus antibody concentration equal or greater than 150 mIU/mL.
Time Frame: At Day 42
Population: ATP cohort for immunogenicity: included all eligible subjects with post-dose serology results available for at least one antigen of measles, mumps, or rubella, who complied with the protocol, who did not meet any elimination criteria and had no intercurrent medical conditions leading to elimination up to the Visit 2 (Day 42) blood sample.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 433 | 436
mIU/mL | 1795.6 [1641.1 to 1964.7] | 1783.3 [1624.6 to 1957.4]
Statistical Analysis 1: Comparison: INV_MMR Group vs COM_MMR Group; Non-inferiority of INV_MMR vaccine to COM_MMR vaccine in terms of Geometric Mean Concentration (GMCs) for anti measles, anti mumps and anti rubella antibodies at Day 42.The 95% CI for adjusted geometric mean concentrations (GMCs) and the adjusted GMC ratio were obtained using an ANCOVA model on the logarithm-transformed concentrations including the vaccine group (for adjusted GMC ratio) as fixed effect, gender, age and country groups as continuous effects and the pre-vaccination log-transformed; Test type: Non-Inferiority or Equivalence — Criteria for the determination of non-inferiority for measles, mumps, and rubella viruses: Lower limit (LL) of the 2-sided 95% Confidence Interval (CI) on GMC ratio (INV_MMR over COM_MMR) was to be equal to or above 0.67 for anti-measles, anti-mumps, and anti rubella antibodies; Adjusted GMC ratio = 1.00, 95% CI 2-sided [0.91 to 1.11] — Number of subjects in the INV-MMR Group and in the COM-MMR Group considered for calculating the adjusted GMC ratio, are respectively 432 and 435 and adjusted GMCs = 1790.2 (LL=1669.6;UL=1919.5) and 1781.5 (LL=1661.8;UL=1909.7) respectively

2. Primary Outcome: Anti-mumps Virus Antibody Concentrations
Description: Antibody concentrations are expressed as Geometric Mean Concentrations (GMCs) in EU/mL. Seropositivity was defined as subjects with anti-mumps virus antibody concentration equal or greater than 5 EU/mL
Time Frame: At Day 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 433 | 436
EU/mL | 110.6 [102.1 to 119.8] | 110.2 [101.9 to 119.2]
Statistical Analysis 1: Comparison: INV_MMR Group vs COM_MMR Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Adjusted GMC ratio = 1.05, 95% CI 2-sided [0.96 to 1.16] — Number of subjects in the INV-MMR Group and in the COM-MMR Group considered for calculating the adjusted GMC ratio, are respectively 432 and 435 and adjusted GMCs = 113.5 (LL=106.0;UL=121.6) and 107.8 (LL=100.7;UL=115.4) respectively

3. Primary Outcome: Anti-rubella Virus Antibody Concentrations.
Description: Antibody concentrations are expressed as Geometric Mean Concentrations (GMCs) in IU/mL. Seropositivity was defined as subjects with anti-rubella virus antibody concentration equal or greater than 4 IU/mL
Time Frame: At Day 42
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: IU/mL
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 433 | 436
IU/mL | 75.3 [70.3 to 80.6] | 75.6 [70.8 to 80.7]
Statistical Analysis 1: Comparison: INV_MMR Group vs COM_MMR Group; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Adjusted GMC ratio = 1.02, 95% CI 2-sided [0.93 to 1.11] — Number of subjects in the INV-MMR Group and in the COM-MMR Group considered for calculating the adjusted GMC ratio, are respectively 432 and 435 and adjusted GMCs = 76.1 (LL=71.5;UL=81.0) and 74.6 (LL=70.2;UL=79.4) respectively

4. Secondary Outcome: Number of Subjects With Anti-measles Virus Antibody Concentration Equal to or Above the Threshold of 200 mIU/mL (Seroresponse Rate)
Description: Seroresponse was defined as:
  Anti-measles virus antibody concentration equal to or above the threshold of 200 mIU/mL after administration of INV_MMR vaccine vs. COM_MMR at Day 42.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 433 | 436
Subjects | 428 | 432

5. Secondary Outcome: Number of Subjects With Anti-mumps Virus Antibody Concentration Equal or Above the Threshold of 10 EU/mL (Seroresponse Rate).
Description: Seroresponse was defined as:
  Anti-mumps virus antibody concentration equal to or above the threshold of 10 EU/mL after administration of INV_MMR vaccine vs. COM_MMR at Day 42.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 433 | 436
Subjects | 426 | 434

6. Secondary Outcome: Number of Subjects With Anti-rubella Virus Antibody Concentration Equal or Above the Threshold of 10 IU/mL (Seroresponse Rate).
Description: Seroresponse was defined as:
  Anti-rubella virus antibody concentration equal to or above the threshold of 10 IU/mL after administration of INV_MMR vaccine vs. COM_MMR at Day 42.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 433 | 436
Subjects | 431 | 435

7. Secondary Outcome: Number of Subjects Who Achieved a 4-fold or Greater Rise in Anti-measles, Anti-mumps and Anti-rubella Virus Antibody Concentrations.
Description: For subjects with seronegative status at pre-vaccination, a 4-fold rise in antibody concentration is defined as 4 times the cut-off level of the assay. Cut-off levels for anti-measles, anti-mumps and anti-rubella virus antibody concentrations are 150 mIU/mL, 5 EU/mL and 4 IU/mL.
Time Frame: At Day 42
Population: as for outcome 1
Measure: Number; unit: Subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 432 | 435
Subjects
  Anti-measles | 42 | 48
  Anti-mumps | 152 | 128
  Anti-rubella | 179 | 161

8. Secondary Outcome: Number of Subjects With Solicited Local Symptoms
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = Occurrence of any local symptom regardless of their intensity grade. Grade 3 Pain = Significant pain at rest. Prevented normal every day activities. Grade 3 redness = redness with surface diameter >50mm. Grade 3 swelling = swelling with surface diameter >50mm.
Time Frame: During the 4-day (Days 0-3) post-vaccination period
Population: Total Vaccinated cohort included all vaccinated subjects with a documented vaccine administration.
Measure: Number; unit: Subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 433 | 445
Subjects
  Any injection site redness | 53 | 52
  Grade 3 injection site redness | 0 | 0
  Any injection site swelling | 23 | 29
  Grade 3 injection site swelling | 0 | 0
  Any injection site pain | 51 | 51
  Grade 3 injection site pain | 1 | 0

9. Secondary Outcome: Number of Subjects Reporting Fever
Description: Fever was assessed:Any fever (≥38°C) = occurrence of any fever regardless of its intensity grade or relationship to vaccination. Grade3 fever = fever >39.5°C. . Related = symptom assessed by the investigator as causally related to study vaccination.The preferred route for recording temperature in this study was oral.
Time Frame: During the 43 days (Days 0-42) post-vaccination period.
Population: Total Vaccinated cohort included all vaccinated subjects with a documented vaccine administration.
Measure: Number; unit: Subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 431 | 445
Subjects
  Any | 13 | 23
  Grade 3 | 1 | 6
  Related | 2 | 6

10. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms as Parotid/Salivary Gland Swelling and Any Sign of Meningism/Seizure.
Description: Assessed MMR specific symptoms were parotid/salivary gland swelling and any sign of meningism/seizure. Parotid/salivary gland swelling: Any = occurrence of any general symptoms regardless of their intensity grade or relationship to vaccination; Grade 3 Parotid/salivary gland swelling = Swelling accompanied with general symptoms. Meningism/seizure: Any= occurrence of any general symptoms regardless of their intensity grade or relationship to vaccination; Grade-3 meningism/seizure= Prevented normal, everyday activities (In adults/adolescents, such an AE could, for example, prevented attendance at work/school and could necessitated the administration of corrective therapy). Related symptom = symptom assessed by the investigator as causally related to study vaccination.
Time Frame: During the 43 days (Days 0-42) post-vaccination period.
Population: Total Vaccinated cohort included all vaccinated subjects with a documented vaccine administration.
Measure: Number; unit: Subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 431 | 445
Subjects
  Any parotid/salivary gland swelling | 1 | 1
  Grade 3 parotid/salivary gland swelling | 1 | 0
  Related parotid/salivary gland swelling | 0 | 0
  Any meningism/seizure | 1 | 1
  Grade 3 meningism/seizure | 1 | 0
  Related meningism/seizure | 0 | 0

11. Secondary Outcome: Number of Subjects Reporting Unsolicited AEs
Description: Any untoward medical occurrence in a patient or clinical investigation child, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product
Time Frame: During the 43 days (Days 0-42) post-vaccination period.
Population: Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 454 | 457
Subjects | 95 | 82

12. Secondary Outcome: Number of Subjects Reporting Solicited Rash Symptom
Description: Assessed any rash, Grade 3, Related, Localized rash, Generalized rash,measles/rubella-rash. Any= occurrence of any general symptom regardless of its intensity grade or relationship to vaccination. Grade3 rash/exanthema= Rash which prevented normal, everyday activities (In adults/adolescents, such an AE could, for example, prevented attendance at work/school and could necessitated the administration of corrective therapy). Grade 3 measles/rubella/varicella-like rash = Rash with more than150 lesions. Related = symptom assessed by the investigator as causally related to study vaccination.
Time Frame: During the 43 days (Days 0-42) post-vaccination period.
Population: Total Vaccinated cohort included all vaccinated subjects with a documented vaccine administration.
Measure: Number; unit: Subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 431 | 445
Subjects
  Any | 9 | 5
  Grade 3 | 0 | 0
  Related | 6 | 2
  Localized rash | 8 | 3
  Generalized rash | 1 | 2
  Rash type - measles/rubella-rash | 0 | 2
  Rash type - others | 9 | 3

13. Secondary Outcome: Number of Subjects Reporting Solicited Joint Pain (Arthralgia/Arthritis)
Description: Assessed any, Grade-3, Related. Any= occurrence of any general symptom regardless of its intensity grade or relationship to vaccination; Grade3 joint pain (arthralgia/arthritis)= Pain which prevented normal, everyday activities (In adults/adolescents, such an AE could, for example, prevented attendance at work/school and could necessitated the administration of corrective therapy). Related = symptom assessed by the investigator as causally related to study vaccination.
Time Frame: During the 43 days (Days 0-42) post-vaccination period.
Population: Total Vaccinated cohort included all vaccinated subjects with a documented vaccine administration.
Measure: Number; unit: subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 431 | 445
subjects
  Any | 8 | 4
  Grade 3 | 0 | 0
  Related | 3 | 1

14. Secondary Outcome: Number of Subjects Reporting NOCDs
Description: Occurrence of new onset chronic diseases (NOCDs)
Time Frame: Day 0 through the end of the study (Day 180)
Population: Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 454 | 457
Subjects | 2 | 1

15. Secondary Outcome: Number of Subjects Reporting Adverse Events Prompting ER Visits
Description: Occurrence of AEs prompting emergency room (ER) visits.
Time Frame: Day 0 through the end of the study (Day 180)
Population: Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 454 | 457
Subjects | 14 | 9

16. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: A serious adverse event (SAE) is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization or results in disability/incapacity.
Time Frame: Day 0 through the end of the study (Day 180)
Population: Total Vaccinated cohort included all vaccinated subjects.
Measure: Number; unit: Subjects
Arm/Group | INV_MMR Group | COM_MMR Group
Number analyzed (Participants) | 454 | 457
Subjects | 3 | 7

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From Day 0 to Day 180, Solicited Local Adverse Events: From Day 0 to Day 3, Solicited General and Unsolicited Adverse Events: From Day 0 to Day 42
Arm/Group | INV_MMR Group | COM_MMR Group
Serious Adverse Events (participants affected / at risk) | 3/454 | 7/457
Other Adverse Events (participants affected / at risk) | 93/454 | 102/457
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INV_MMR Group (N=454) | COM_MMR Group (N=457)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis relapsing (Gastrointestinal disorders) | 0 (0) | 1 (1)
Biliary colic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2)
Psychogenic seizure (Psychiatric disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | INV_MMR Group (N=454) | COM_MMR Group (N=457)
Injection site erythema (General disorders) | 53 (53) | 52 (52)
Injection site swelling (General disorders) | 23 (23) | 29 (29)
Pyrexia (General disorders) | 13 (13) | 23 (23)
Vaccination site pain (General disorders) | 51 (51) | 51 (51)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.